CLINICAL TRIAL: NCT01515592
Title: A Randomised, Double-blind Within Dose Group, Single Centre, Placebo-controlled, Dose Escalation, Multiple s.c. Dose Study to Assess the Safety and Tolerability of Liraglutide 20 ug/kg and 25 ug/kg in Healthy Japanese Male Subjects
Brief Title: Safety and Tolerability of Liraglutide in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1694
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- 20 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- 25 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — One daily subcutaneous dose for 5 weeks. Dose is weekly incremented with 5 mcg/kg
  Arms: 15 mcg/kg
Drug: liraglutide — One daily subcutaneous dose for 5 weeks. 5 mcg/kg the first week, then 10 mcg the second week followed by 15 mcg the third week, and finally 20 mcg for 2 weeks
  Arms: 20 mcg/kg
Drug: liraglutide — One daily subcutaneous dose for 5 weeks. 5 mcg/kg the first week, then 10 mcg the second week followed by 15 mcg for 3 weeks
  Arms: 25 mcg/kg
Drug: placebo — Liraglutide placebo administered to subjects randomised at each dose level in the ratio of 3:1

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to assess the safety and tolerability of 20 µg/kg and 25 µg/kg liraglutide in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects
* BMI (Body Mass Index) between 18.0-27.0 kg/m^2 inclusive

Exclusion Criteria:

* Any clinical laboratory values deviated from the reference range at the laboratory (except for cases within physiological change) or any abnormal ECG (electrocardiogram) findings at the screening
* Presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies positive
* History of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* History of significant allergy or hypersensitivity
* Known or suspected allergy to trial product or related products
* History of drug or alcohol abuse
* The subjects who smoke more than 15 cigarettes, or the equivalent, per day and is unwilling to refrain from smoking whenever required for the trial procedure

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Adverse events
Body weight
Antibody against liraglutide

SECONDARY OUTCOMES:
Area under the plasma liraglutide concentration curve
Cmax, maximum concentration
tmax, time to reach Cmax
Terminal elimination rate constant
t½, terminal elimination half-life
24-hour profiles of plasma glucose
24-hour profiles of serum insulin

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Irie S, Matsumura Y, Zdravkovic M, Jacobsen LV, Kageyama S. Tolerability, pharmacokinetics and pharmacodynamics of the once-daily human GLP-1 analog liraglutide in Japanese healthy subjects: a randomized, double-blind, placebo-controlled dose-escalation study. Int J Clin Pharmacol Ther. 2008 Jun;46(6):273-9. doi: 10.5414/cpp46273. PMID 18541123
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com